CLINICAL TRIAL: NCT01426022
Title: The Effect of Moderate Alcohol Consumption With a Meal in Different Ambiances on Postprandial Mood, Evaluated by Subjective and Physiological Responses
Brief Title: Effect of Moderate Alcohol Consumption on Postprandial Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Responsible Party: Principal Investigator, Henk FJ Hendriks, PhD, TNO
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: P9334
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Mood Swings
Keywords: alcohol; mood; postprandial
MeSH Terms: interventions — Nutritional Status; Ethanol; Wine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol (Placebo Comparator): 1. 3 glasses of sparkling white wine (30g alcohol) with dinner
  2. 3 glasses of alcohol free sparkling white wine (<2g alcohol) with dinner
  Interventions: Other: Nutrition
- Ambiance (Experimental): 1. Pleasant ambiance
  2. Unpleasant ambiance
  Interventions: Behavioral: mood manipulation

INTERVENTIONS:
Other: Nutrition — Moderate alcohol consumption with dinner (3 glasses of sparkling white wine, containing ca. 30 g alcohol)
  Other Names: Alcohol; Ethanol; Wine
  Arms: Alcohol
Behavioral: mood manipulation — Mood will be manipulated by changing the ambiance in either a pleasant or unpleasant way.
  Other Names: Ambience; Ambiance; Positive affect; Emotion
  Arms: Ambiance

SUMMARY:
Rationale: Food choice is influenced by postprandial mood; the feelings of well-being after a meal. Postprandial mood can be measured by subjective responses. Physiological responses may play an important role in the generation of postprandial mood. However, the relationship between subjective and physiological responses after a meal is not clear yet. To investigate this relationship, moderate alcohol consumption will be used as a mood modulator, because of its well-studied effects on mood. Postprandial mood depends on the current mood state. Therefore the investigators will manipulate the current mood state by changing the ambiance to measure the influence of moderate alcohol consumption with a meal on postprandial mood in a pleasant or unpleasant ambiance.

Objective: To determine whether moderate alcohol consumption with a meal in different ambiances affects postprandial mood, evaluated by subjective and physiological parameters.

Study design: Randomized, placebo-controlled, single-blind, cross-over trial

Study population: 28 apparently healthy, normal weight (BMI 18.5-27 kg/m2) women (18-45 y), taking oral contraceptives.

Intervention: 4 times having dinner at TNO Zeist with either 3 glasses of sparkling white wine (~30g alcohol) or alcohol-free sparkling white wine in either a pleasant or unpleasant meal ambiance.

Hypothesis: It is hypothesized that moderate alcohol consumption with a meal in different ambiances changes the response of subjective and physiological parameters of mood.

* Ho: there is no effect of alcohol consumption and ambiance on mood
* H1: there is an effect of alcohol consumption and ambiance on mood

ELIGIBILITY:
Inclusion Criteria:

* Healthy as assessed by the health and lifestyle questionnaire, (P9334 F02; in Dutch)
* Females aged 18-45 years at Day 01 of the study
* Taking a monophasic combined oral contraceptive pill at Day 01 of the study, with 21 days of taking pills with active ingredients followed by 7 days taking no pills or continuous intake of the oral contraceptive pill
* Body Mass Index (BMI) of 18.5-27 kg/m2
* Body weight between 57 and 80 kg
* Normal Dutch eating habits as assessed by P9334 F02
* Alcohol consumption ≥ 3 and ≤ 21 standard units/week
* Voluntary participation
* Having given written informed consent
* Willing to comply with the study procedures, including refrain from alcohol 24 h before the test days and refrain from caffeine during the afternoon of the test day
* Appropriate veins for blood sampling/cannula insertion according to TNO
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
* Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study.
* Having a history of medical or surgical events or disease that may significantly affect the study outcome, particularly physiological disorders, or psychiatric, metabolic or endocrine disease and gastrointestinal disorders.
* Use of medication that may affect the outcome of the study parameters (e.g. antidepressive drugs).
* Having a family history of alcoholism
* Having a history of alcohol or drug related problems
* Smoking
* Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
* Reported slimming or medically prescribed diet
* Reported vegan, vegetarian or macrobiotic
* Recent blood donation (<1 month prior to the start of the study)
* Not willing to give up blood donation during the study.
* Pregnant (to their own knowledge) or lactating or wishing to become pregnant in the period of the study
* Personnel of TNO Zeist, their partner and their first and second degree relatives
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Profile of mood states (POMS) | 5 times during study day, 4 study days (total 20x)
  Difference between the change in the score of the 6 items of the POMS (after consumption of either white wine or alcohol free white wine with a meal in either a positive or negative ambiance. POMS will be measured before consumption, and 30min, 60min, 90min and 150min after consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Henk Hendriks, PhD, Principal Investigator — TNO
Locations (1):
- TNO, Zeist, Utrecht, Netherlands

REFERENCES:
- [Derived] Schrieks IC, Ripken D, Stafleu A, Witkamp RF, Hendriks HF. Effects of mood inductions by meal ambiance and moderate alcohol consumption on endocannabinoids and N-acylethanolamines in humans: a randomized crossover trial. PLoS One. 2015 May 11;10(5):e0126421. doi: 10.1371/journal.pone.0126421. eCollection 2015. PMID 25962070
- [Derived] Schrieks IC, Stafleu A, Kallen VL, Grootjen M, Witkamp RF, Hendriks HF. The biphasic effects of moderate alcohol consumption with a meal on ambiance-induced mood and autonomic nervous system balance: a randomized crossover trial. PLoS One. 2014 Jan 21;9(1):e86199. doi: 10.1371/journal.pone.0086199. eCollection 2014. PMID 24465955